CLINICAL TRIAL: NCT04266977
Title: Restrictive Use of Dexamethasone in Glioblastoma
Acronym: RESDEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RESDEX
Record Dates: First submitted 2020-02-03; First posted 2020-02-12 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Glioblastoma; Dexamethasone; Steroids
MeSH Terms: conditions — Glioblastoma | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: restrictive use of DEX, based on standardized clinical and radiological criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Dexamethasone (Experimental): The restrictive DEX regimen is applied from referral to the neurosurgical center until discharge. All administered steroids will be stopped immediately after study inclusion.
  If one or more of the previously defined failure criteria occurs, patients will be treated with DEX.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — restrictive use of DEX, based on standardized clinical and radiological criteria.

SUMMARY:
The administration of steroids, most commonly dexamethasone (DEX), has established as standard of care during treatment of glioblastoma (GBM) and is widely used during the entire course of the disease including pre- and postoperative management, chemo- and radiotherapy. The primary purpose is to reduce tumor-associated vasogenic edema and to prevent or treat increased intracranial pressure. However, steroids are also linked to a multitude of adverse side effects that may affect survival of GBM patients such as major immunosuppression. The use of steroids during radiotherapy is associated with reduced overall- and progression-free survival and has been identified as an independent poor prognostic factor. Despite these findings, the suspicion of GBM often triggers the administration of DEX in routine clinical practice, regardless of neurological symptoms, tumor size, or extension of cerebral edema. The purpose of this study is to assess whether selected GBM patients can be treated safely with a restrictive DEX regimen from referral to the neurosurgical center until discharge.

The primary objective is to determine the failure rate of a restrictive DEX regimen defined as edema or mass effect leading to any of the following: GCS deterioration ≥ 2 points, NIHSS increase ≥ 3 points, increase of midline Shift ≥ 2mm, or any surgical rescue procedure for increasing mass effect.

DETAILED DESCRIPTION:
Background

Glioblastoma (GBM) is the most common and devastating malignant brain tumor in adults. Patients with glioblastoma face a poor prognosis. Despite maximal treatment, most patients suffer tumor progression after 6-7 months and die within 1-2 years. Standard treatment for newly diagnosed glioblastoma contains maximal safe surgery and adjuvant radiochemotherapy with temozolomide. Additional administration of steroids has established as standard of care during treatment of GBM. It is widely used during the entire course of the disease including pre- and postoperative management, chemotherapy and radiotherapy. Dexamethasone (DEX) is the most frequently used steroid. The main purpose is to reduce the tumor associated vasogenic cerebral edema, to prevent or treat increased intracranial pressure. In addition, DEX helps to cope with adverse effects of GBM-treatment like nausea, vomiting and fatigue. However, steroids are also linked to a multitude of adverse side effects that may affect the survival of GBM patients such as major immunosuppression, and metabolic changes like hyperglycemia. The use of steroids during radiotherapy is associated with reduced overall- and progression-free survival and has been identified as an independent poor prognostic factor. DEX was also related to a poor prognosis in recurrent GBM. Despite these findings, in routine clinical practice, the suspicion of glioblastoma often triggers the administration of DEX, regardless of neurologic symptoms or the extension of cerebral edema. Many patients are treated with larger doses of DEX per day before being referred to a neurosurgical center and are kept on steroids during the entire treatment. On the other hand, the clinical experience shows that GBM-patients with no, or only mild neurologic symptoms, normal intracranial pressure and relatively small cerebral edema can be managed without administration of DEX. The rationale for this study is to objectify the criteria and safety of a restrictive DEX regimen (based on standardized clinical and radiological criteria). A restrictive DEX regimen may help to reduce over-use, limit the number of patients exposed to the adverse effects of DEX, and potentially improve survival in GBM-patients. The purpose of this study is to assess whether selected GBM patients can be treated safely with a restrictive DEX regimen from referral to the neurosurgical center until discharge.

Objective

The primary objective is to determine the failure rate of a restrictive DEX regimen defined as edema or mass effect leading to any of the following: GCS deterioration ≥ 2 points, NIHSS increase ≥ 3 points, increase of midline Shift ≥ 2mm, or any surgical rescue procedure for increasing mass effect.

Methods

All patients referred to the neurosurgical center with suspicion of glioblastoma are screened for inclusion- and exclusion criteria. If eligible and consenting of the patient to the study protocol, no steroids will be administered until discharge (except optional intraoperative single shot dexamethasone of max. 4mg if necessary). If steroids have been administered for a maximum of one day before referral, they will be stopped immediately. Patients are followed clinically. If one of the above-described failure criteria occurs, the primary endpoint is reached and DEX will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed supratentorial contrast enhancing lesion suspicious of glioblastoma without major mass effect, amenable to surgical resection
* Age 18 - 90 years
* Midline Shift ≤ 3mm
* GCS ≥ 14
* NIHSS ≤ 3
* Provided written informed consent

Exclusion Criteria:

* Infratentorial lesions, brainstem lesions, multifocal lesions
* Therapy with steroids for >1 day before inclusion
* Need for treatment with steroids due to any other disease
* Contraindications to the administration of Dexamethasone
* Pregnancy or breastfeeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-05-08 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Failure rate of the restrictive DEX regimen | 30 days after surgery
  Failure rate of the restrictive DEX regimen, defined as cerebral edema or mass effect causing any of the following: GCS deterioration ≥ 2 points or NIHSS increase ≥ 3 points or Increase of midline Shift ≥ 2mm or any new herniation sign on imaging or Any surgical rescue procedure for increasing mass effect (hemicraniectomy, removal of bone flap, abortion of the procedure or emergency tumor debulking

SECONDARY OUTCOMES:
Secondary neurological or systemic complication | 30 days after surgery
  Secondary neurological or systemic complication resulting in a 30-day morbidity or mortality
Cumulative dexamethasone dosage | 30 days after surgery
  Cumulative dexamethasone dosage during study period
National Institutes of Health Stroke Scale (NIHSS) over time of the study period | 30 days after surgery
  NIHSS over time of the study period and correlation with steroid medication (Score 0-42, 0 = no deficits and 1-42 deficits)
Glasgow Coma Scale (GCS) over time of the study period and correlation with steroid medication | 30 days after surgery
  GCS over time of the study period and correlation with steroid medication GCS over time of the study period and correlation with steroid medication (Score 15-3, 15 = patient is fully oriented, 3 = patient is intubated)
Volume of contrast enhancing tumor on preoperative MRI | presurgery
  Volume of contrast enhancing tumor on preoperative MRI
Volume of contrast enhancing tumor on postoperative MRI | 48 hours after surgery
  Volume of contrast enhancing tumor on postoperative MRI
Volume of edema on preoperative MRI and correlation with steroid medication | presurgery
  Volume of edema on preoperative MRI and correlation with steroid medication
Volume of edema on postoperative MRI | 48 hours after surgery
  Volume of edema on postoperative MRI and correlation with steroid medication
Time to start of adjuvant treatment | 30 days after surgery
  Time to start of adjuvant treatment
Rate of reoperations | 30 days after surgery
  Rate of reoperations
Cause of reoperations | 30 days after surgery
  Cause of reoperations

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Raabe, MD, Principal Investigator — Inselspital Bern, Department of Neurosurgery
Locations (4):
- Switzerland (4):
  - Kantonsspital St. Gallen, Sankt Gallen, St.Gallen
  - Universitätsspital Basel, Basel
  - Department of Neurosurgery, Bern
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] GALICICH JH, FRENCH LA, MELBY JC. Use of dexamethasone in treatment of cerebral edema associated with brain tumors. J Lancet. 1961 Feb;81:46-53. No abstract available. PMID 13703072
- [Background] KOFMAN S, GARVIN JS, NAGAMANI D, TAYLOR SG 3rd. Treatment of cerebral metastases from breast carcinoma with prednisolone. J Am Med Assoc. 1957 Apr 20;163(16):1473-6. doi: 10.1001/jama.1957.02970510039008. No abstract available. PMID 13415910
- [Background] Luedi MM, Singh SK, Mosley JC, Hassan ISA, Hatami M, Gumin J, Andereggen L, Sulman EP, Lang FF, Stueber F, Fuller GN, Colen RR, Zinn PO. Dexamethasone-mediated oncogenicity in vitro and in an animal model of glioblastoma. J Neurosurg. 2018 Dec 1;129(6):1446-1455. doi: 10.3171/2017.7.JNS17668. Epub 2018 Jan 12. PMID 29328002
- [Background] Ly KI, Wen PY. Clinical Relevance of Steroid Use in Neuro-Oncology. Curr Neurol Neurosci Rep. 2017 Jan;17(1):5. doi: 10.1007/s11910-017-0713-6. PMID 28138871
- [Background] Pitter KL, Tamagno I, Alikhanyan K, Hosni-Ahmed A, Pattwell SS, Donnola S, Dai C, Ozawa T, Chang M, Chan TA, Beal K, Bishop AJ, Barker CA, Jones TS, Hentschel B, Gorlia T, Schlegel U, Stupp R, Weller M, Holland EC, Hambardzumyan D. Corticosteroids compromise survival in glioblastoma. Brain. 2016 May;139(Pt 5):1458-71. doi: 10.1093/brain/aww046. Epub 2016 Mar 28. PMID 27020328
- [Background] Roth P, Wick W, Weller M. Steroids in neurooncology: actions, indications, side-effects. Curr Opin Neurol. 2010 Dec;23(6):597-602. doi: 10.1097/WCO.0b013e32833e5a5d. PMID 20962642
- [Background] Shields LB, Shelton BJ, Shearer AJ, Chen L, Sun DA, Parsons S, Bourne TD, LaRocca R, Spalding AC. Dexamethasone administration during definitive radiation and temozolomide renders a poor prognosis in a retrospective analysis of newly diagnosed glioblastoma patients. Radiat Oncol. 2015 Oct 31;10:222. doi: 10.1186/s13014-015-0527-0. PMID 26520780
- [Background] Ueda S, Mineta T, Nakahara Y, Okamoto H, Shiraishi T, Tabuchi K. Induction of the DNA repair gene O6-methylguanine-DNA methyltransferase by dexamethasone in glioblastomas. J Neurosurg. 2004 Oct;101(4):659-63. doi: 10.3171/jns.2004.101.4.0659. PMID 15481722
- [Background] Wong ET, Lok E, Gautam S, Swanson KD. Dexamethasone exerts profound immunologic interference on treatment efficacy for recurrent glioblastoma. Br J Cancer. 2015 Dec 1;113(11):1642. doi: 10.1038/bjc.2015.404. No abstract available. PMID 26625224
- [Background] Weinstein JD, Toy FJ, Jaffe ME, Goldberg HI. The effect of dexamethasone on brain edema in patients with metastatic brain tumors. Neurology. 1973 Feb;23(2):121-9. doi: 10.1212/wnl.23.2.121. No abstract available. PMID 4734508
- [Result] Derr RL, Ye X, Islas MU, Desideri S, Saudek CD, Grossman SA. Association between hyperglycemia and survival in patients with newly diagnosed glioblastoma. J Clin Oncol. 2009 Mar 1;27(7):1082-6. doi: 10.1200/JCO.2008.19.1098. Epub 2009 Jan 12. PMID 19139429